CLINICAL TRIAL: NCT03075930
Title: A Registry With the Aim to Identify Characteristics of Atrial Conduction and Risk of Recurrence in Patients With Atrial Fibrillation Undergoing Ablation for Atrial Fibrillation
Brief Title: Atrial Fibrillation Ablation Registry
Acronym: AFAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Matthias D Zink, Principal Investigator, Maastricht University Medical Center
Other Study IDs: METC 16-4-208
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation (Paroxysmal); Atrial Fibrillation Recurrent; Atrial Fibrillation Common Gene Variants
Keywords: Atrial fibrillation; ECG; Body surface potential map; Recurrence of AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Probes of blood for common gene variant analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extended Electrocardiogram: Elective patients receiving an AF ablation receiving a extended ECG
  Interventions: Device: Extended Electrocardiogram
- Body surface potential map: Elective patients receiving an AF ablation receiving a body surface potential map
  Interventions: Device: Body surface potential map

INTERVENTIONS:
Device: Extended Electrocardiogram — ECG with 3 additional leads and a 5 minute recording
  Groups: Extended Electrocardiogram
Device: Body surface potential map — ECG with 184 leads and a 5 minute recording
  Groups: Body surface potential map

SUMMARY:
This is a single centre prospective data registry. In this study atrial conduction characteristics of extended surface Electrocardiograms (esECG), biomarkers and genetic analysis will be performed before ablation, before discharge and 3 months after catheter ablation of atrial fibrillation (AF) and compared to routine clinical follow-up data.

The objective of this registry is to establish a data registry of patients undergoing ablation of AF. Supplementary to the routine clinical diagnostic an esECG and an analysis of biomarkers will be performed and compared to clinical and outcome data.

DETAILED DESCRIPTION:
Electro anatomical remodelling of the atria due to ageing or structural heart disease leads to AF which in turn leads to cardiac electrical and structural remodelling. In case of advanced remodelling restoration of sinus rhythm (SR) becomes more difficult and the results of catheter ablation are disappointing. Furthermore, there is no valid parameter to predict or diagnose recurrence of AF during SR after successful ablation, so repeated long-term electrocardiogram (ECG) recordings have to be performed to detect asymptomatic AF episodes in particular.

Thus, the rationale to establish a systematic review of patient data in a registry are:

* Self-termination AF leads to slight, persistent AF leads to more advanced cardiac remodelling, shown in altered atrial conduction properties
* Early recognition and therapy of AF improves the outcome, thus clinical parameter to predict or diagnose recurrence of AF during SR are desirable Ablation of AF is predominantely performed using standard endocardial transvenous technique of pulmonary veins isolation (PVI) by radiofrequency or cryoballoon ablation. For medical reasons specific ablation techniques like additional ablation lines or an epicardial approach is in discretion of the treating cardiologist. The esECG is measured by signal averaged routine 12-lead ECG with 3-5 supplementary leads before ablation, before discharge and 3 months after ablation. 2 tubes of EDTA plasma will be taken supplementary during routine venous puncture on admission and analysed for biomarkers and common gene variants.

During 5 years every participant receives an esECG before ablation, before discharge and three months after ablation. Routine follow-up data of each participant is included until 12 months of follow-up.

Patients who are included would also undergo a procedure without participation in this study. Risks (complications of procedures) are associated with the procedure and not with participation in the registry. The supplementary diagnostics performed for the registry are comprehensible to clinical routine ECG diagnostics. Extra (study-related) investigations consist of esECG (a signal averaged surface ECG with 3-5 supplementary leads at baseline before ablation), before discharge, and 3 months after ablation, and possibly also a body surface potential map (BSPM). These are always planned together with routine follow-up, no extra visits are necessary. The esECG and BSPM can be compared to regular ECGs, the only additional discomfort might be the number of leads. Furthermore 2 tubes of EDTA plasma blood will be taken supplementary at the routine admission venous puncture for further biomarker and common gene variants analysis.

Quality assurance plan: All data will be stored in 2 independent database. In the first database personal and contact informations are stored with a decent patient ID number in ascending order. In the other database all medical informations will be stored without personal data of the patient. The database has algorithm to prevent mesenteries and rudimentary checks for data integrity and consistency. List are provided for repeated parameters and all variables are explained if relevant. Standard operating procedures are provided for relevant steps in patient inclusion, measurements and data entry.

Because of the registry character no sample size calculation is provided yet. But after the first year of inclusion a data analysis will provide informations about an expected sample size. To date we calculate for an period of patient inclusion of 5 years.

Data inconsistency could not be avoided due to the registry character of this study and will marked in a respective way.

Statistical analysis will be performed after the first year of patients including logistic regression analysis to determine the discriminative power of the recorded ECG for the clinical outcome and recurrence of AF.

ELIGIBILITY:
Inclusion Criteria:

* Documented self-terminating or persistent AF
* Scheduled for ablation of AF
* At least 18 years of age, mentally able and willing to give informed consent

Exclusion Criteria:

* Emergency ablation
* Serious patient condition before ablation
* Physically or mentally unable to provide written informed consent
* Permanent atrial fibrillation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for ablation of AF with a history of self-terminating or persistent non-valvular AF with at least one documented AF episode during the last 6 months
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of AF after ablation | 12 months
  The predictive value for recurrence of AF in patients after ablation of AF based on atrial conduction characteristics in electrocardiographic, -anatomical, biomarker and genetic analysis

SECONDARY OUTCOMES:
AF characteristics | 12 months
  Identify characteristics of patients with self-terminating in contrast to patients with persistent AF in the registry data
ECG AF characteristics | 3 months
  Identify changes by ablation and convalescence in the extended surface ECG
ECG to BSPM discriminative power | 12 months
  To compare the registry data with a subgroup analysis receiving additional to the routine diagnostics a body surface potential map (BSPM) and an ECG-Imaging (ECGI)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pison, Physician, Study Director — Maastricht University; Ulrich Schotten, Physician, Principal Investigator — Maastricht University; Matthias D Zink, Physician, Study Director — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
This study is planned as a Single Center Study. But it could be possible to extend it to other centers. In this case data will be shared with the participating centers.
Supporting Information: Study Protocol
Time Frame: In case of an extend to another participating center IPD are available for the collaborating center.
Access Criteria: In case of an extend to another participating center IPD are available for the collaborating center.